CLINICAL TRIAL: NCT00879320
Title: Healthy Lifestyle in Adults With ADHD
Brief Title: Healthy Lifestyle in Adults With Attention Deficit Hyperactivity Disorder
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, Thomas J. Spencer, MD, Associate Chief, Clinical and Research Program, Pediatric Psychopharmacology, Massachusetts General Hospital
Other Study IDs: 2008-P-002056
Record Dates: First submitted 2009-04-09; First posted 2009-04-10 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: ADHD; Attention Deficit Hyperactivity Disorder
Keywords: ADHD; health; healthy lifestyle
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Adults with ADHD
- 2: Healthy adults without ADHD

SUMMARY:
The purpose of this study is to understand the relationship between ADHD and the overall health of someone with ADHD. People who have ADHD have trouble paying attention, concentrating, organizing, and planning. They may have trouble in school, at work, and at home. The investigators are interested in finding out whether these difficulties have had any influence in the past, current, or future health problems of someone with ADHD. About 100 people with ADHD and 100 people without ADHD will take part in this research study, all through Massachusetts General Hospital (MGH).

ELIGIBILITY:
Inclusion Criteria:

ADHD Subjects

1. Signed written informed consent to participate in the study.
2. Age: 18 - 60 (inclusive).
3. Current diagnosis of DSM-IV ADHD by structured interview. Late age of onset acceptable for participation provided ADHD symptoms meet full criteria currently.

Control Subjects

1. Signed written informed consent to participate in the study.
2. Age: 18 - 60 (inclusive).
3. Subjects must have <3 symptoms in each domain (Inattention and Hyperactive/Impulsive) and <5 total symptoms in both domains on the DSM-IVADHD module of the structured interview.

Exclusion Criteria:

1. Diagnosis of any psychotic disorder or Autism.
2. Mental impairment as evidenced by a Full Scale I.Q. less than 80.
3. Major sensorimotor handicaps such as deafness or blindness.
4. Subject currently taking antipsychotic medication or mood stabilizers.
5. Inadequate command of the English language.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adults ages 18-55 who have ADHD (for ADHD group) Healthy adult volunteers ages 18-55 who do not have ADHD (control group)
Sampling Method: Non-Probability Sample
Enrollment: 253 (Actual)
Dates: Start 2009-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Comparison of ADHD and control subject health habits will be assessed by subject-rated questionnaires and health measures, such as vital signs and blood draw results. | 1 time

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Spencer, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States